CLINICAL TRIAL: NCT00650741
Title: Evaluation of a New Non-Invasive Device for Detection of Endothelial Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Lavi Cardiatec (Industry)
Responsible Party: Avner Amir CEO, Lavi Cardiatec
Other Study IDs: SMC0001
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Endothelial Dysfunction
Keywords: Endothelial Dysfunction; FMD

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 10 subjects, Half with Endothelial Dysfucntion (according to previous ultrasound FMD) , Half with no endothelial dysfucntion (according to previous ultrasound FMD), no repetition of test
- 2: 10 subjects, Half with Endothelial Dysfucntion (according to previous ultrasound FMD) , Half with no endothelial dysfucntion (according to previous ultrasound FMD), Repetition with Nitroglycerin
- 3: 10 subjects, Half with Endothelial Dysfucntion (according to previous ultrasound FMD) , Half with no endothelial dysfucntion (according to previous ultrasound FMD), repetition of test with the Endotect

SUMMARY:
The purpose of the study is to investigate the sensitivity and specificity of the Endotect compared with an ultrasound device in a flow-mediated vasodilatation (FMD) test.

DETAILED DESCRIPTION:
The study compares the results obtained with Endotect with the results obtained from a brachial ultrasound FMD test, with and without nitroglycerin.

The results from 3 patient groups (see below) will be compared

1: 10 subjects, Half with Endothelial Dysfucntion (according to previous ultrasound FMD) , Half with no endothelial dysfucntion (according to previous ultrasound FMD), no repetition of test 2: 10 subjects, Half with Endothelial Dysfucntion (according to previous ultrasound FMD) , Half with no endothelial dysfucntion (according to previous ultrasound FMD), Repetition with Nitroglycerin 3: 10 subjects, Half with Endothelial Dysfucntion (according to previous ultrasound FMD) , Half with no endothelial dysfucntion (according to previous ultrasound FMD), repetition of test with the Endotect

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18-65.
2. Ambulatory
3. FMD ultrasound assessment within past 6 months.
4. No clinical evidence of cardiovascular disease (no history of MI, TIA or stroke, limp, carotid or aortic murmurs)
5. 10 hour fast - water only
6. Normal peripheral pulse examination.
7. ECG without evidence of former MI or LVH.
8. Capable of understanding the explanation and signing informed consent.

Exclusion Criteria:

1. Below age 18 and above age 65.
2. Pregnancy
3. Has not had FMD ultrasound assessment within past 6 months.
4. Exhibits clinical evidence of cardiovascular disease (history of MI, TIA or stroke, limp, carotid or aortic murmurs, clotting disorder)
5. Has eaten or drunk anything besides water in past 10 hours.
6. Known sensitivity to NTG
7. Takes medication for asthma, heart disease or depression, such as atenolol (Tenormin); carteolol (Cartrol); labetalol (Normodyne,Trandate); metoprolol (Lopressor); nadolol (Corgard); phenelzine (Nardil); propranolol (Inderal); sotalol (Betapace); theophylline (Theo-Dur); timolol (Blocadren); tranylcypromine (Parnate), and tricyclic antidepressants such as Elavil
8. Anemia, glaucoma, or have taken medication such as calcium channel blockers like amlodipine (Norvasc), diltiazem(Cardizem), felodipine (Plendil), isradipine (DynaCirc), nifedipine (Procardia), and verapamil (Calan, Isoptin); dihydroergotamine (D.H.E. 45)
9. Venopuncture of arms within past week
10. Use of Viagra, Levitra, Cialis or similar medications to treat erectile dysfunction within last 24 hours or planned use within 8 hours
11. Any of the following:

    * unstable emotionally
    * unable to understand explanation of study
    * ECG with evidence of former MI or LVH.
    * Abnormal peripheral pulses
12. Has not signed an informed consent form.
13. Patient is enrolled in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who visited a clinic where FMD is performed and community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-02

CONTACTS AND LOCATIONS:
Overall Officials: Giora Amitzur, Ph. D., Study Director — Heart Institute, Sheba Medical Center and Tel Aviv University, Israel; Michael Schechter, MD MA FACC, Principal Investigator — Heart Institute, Sheba Medical Center, Israel
Locations (1):
- Sheba Medical Center, Heart Institutue, Tel Litwinsky, Israel